CLINICAL TRIAL: NCT01111942
Title: A Pilot Study of Induction Chemotherapy Followed by Surgery for Locally Advanced Resectable Head and Neck Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: Southern Illinois University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ROB-SCCI 10-001-1
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer; chemotherapy; radiation
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Docetaxel; Cisplatin; Fluorouracil; Bloodless Medical and Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- radiation and weekly carboplatin (Active Comparator)
  Interventions: Other: radiation combined with weekly carboplatin
- conservation surgery (Other)
  Interventions: Procedure: conservation surgery

INTERVENTIONS:
Other: radiation combined with weekly carboplatin — recommended premedications: Aloxi 0.25 mg IV; Dexamethasone 20 mg IV; Fosaprepitant 115 mg IV; Aprepitant 80 mg PO; Ativan 1.0 mg IV;
  Mucositis treatment should involve local measures to maintain oral hygiene, oral nystatin or fluconazole, or valacyclovir for viral infection.
  Induction Triple Therapy Treatment with TPF:
  Docetaxel (Taxotere) 75 mg/m2 IV; Cisplatin (Platinol) 100 mg/m2 IV; 1500 cc Normal Saline w/20meq KCL, 1 gram MgSo4 IV; 5-Fluorouracil (Adrucil) 1000 mg/m2 day IV-continuous infusion over 4 days; Neulasta* 6 mg SC Day 5 (*Neupogen may be substituted at the investigator's discretion)
  Other Names: Docetaxel; Taxotere; Cisplatin; Platinol; 5-Fluorouracil; Adrucil
  Arms: radiation and weekly carboplatin
Procedure: conservation surgery — Following induction triple chemotherapy, subjects will be restaged by physical examination and radiological imaging. If there is an absence of unequivocal evidence for residual disease (i.e. an apparent complete response), the subject will undergo conservation surgery under general anesthesia, using a transoral approach. Minimal tissue removal through direct access. The surgical specimen will be evaluated by a pathologist in the manner standard for the institution. The presence of residual tumor will be classified as a partial response to induction triple chemotherapy and the subject will undergo concomitant chemoradiotherapy. If there is no evidence of residual disease in the surgical specimen, the subject will be followed for recurrence.
  Other Names: Docetaxel; Taxotere; Cisplatin; Platinol; 5-Fluorouracil; Adrucil
  Arms: conservation surgery

SUMMARY:
This is a non-randomized open-label investigator initiated pilot study comparing follow-up therapy of advanced head and neck cancer subjects initially treated with triple induction chemotherapy. Subjects will receive surgical treatment or combined chemoradiation therapy based on the subject's apparent clinical response. Spared use of radiation therapy for selective patients who have a complete response to induction chemotherapy could improve well being of this patient population without compromising survival.

DETAILED DESCRIPTION:
An important observation of the induction triple chemotherapy regimen know as TPF is that there was an unprecedented high proportion of patients treated who had a complete response of their disease upon the completion of the induction phase. In a recent study by Haddad, et al., a biopsy was performed in all patients following induction chemotherapy and before starting concomitant chemoradiotherapy. Patients with an incomplete response to chemoradiotherapy or who had N3 disease had a neck dissection 6 to 12 weeks after chemoradiotherapy. Twenty-nine neck dissections were performed after chemoradiotherapy. The neck dissection result was pathologically positive in 7 (24%) patients (all alive with no evidence of disease) and negative in 22 (76%) patients (21 alive with no evidence of disease). Post-TPF, primary site biopsy result was negative in 64 patients (89%) and positive in 8 patients (11%). While the protocol required all patients to subsequently receive concomitant chemoradiation regardless of disease response to the induction component of the regimen, it is reasonable to question whether the complete responder subset really needed to undergo the same intensive chemoradiation treatment compared to the partial responders. Thus, a less intense therapy may be sufficient. The long term goal of this protocol is to alter the model of highly effective cancer therapy from what is maximally tolerated by the patient to what is minimally necessary for a cure.

One treatment strategy for patients with advanced head and neck cancer who prove to be highly sensitive to chemotherapy is to combine the modalities of polychemotherapy and conservation surgery with the goal of avoiding radiation therapy. For those patients whose primary disease is classified as T2-3 (resectable), and who have a complete response following induction therapy, it is feasible to perform an organ preservation tumor nidusectomy at the primary site to verify that the clinical complete response is truly pathological complete response. Similarly, the clinical complete response observed for the associated nodal disease, can be verified pathologically by performing a selective neck dissection without causing significant morbidity. Both tumor nidusectomy and selective neck dissection has been shown to be an effective adjuvant in this setting. Building on these observations, the novel protocol outlined in this proposal has the potential to spare the use of radiation therapy for selective patients who have a complete response to induction chemotherapy and thereby improve their well being without compromising survival.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent document.
2. Histologically confirmed Stage III-IV (T1, T2, T3) (N0-N2) squamous cell carcinoma of the oropharynx staged according to AJCC guidelines.
3. The subject must be considered surgically resectable via a transoral approach at the time of presentation.
4. Age >18 years
5. Life expectancy >/= 5 years
6. ECOG performance status <2
7. Subject must have measurable disease, at least one lesion accurately measured in at least one dimension as >10 mm with CT scan.
8. Hematologic Absolute neutrophil count > 1,000/mm3, Hemoglobin > 8.0 g/dl Platelet count > 100,000/mm3 Leukocytes >3,000/mcL
9. Hepatic Total Bilirubin ≤ ULN; AST and ALT and Alkaline Phosphatase within the eligible range
10. Renal - creatinine within normal institutional limits or >60 mL/min/1.73 m2 creatinine > institutional normal
11. Women of childbearing potential with negative pregnancy test.
12. Men and women of childbearing age willing to use effective contraception

Exclusion Criteria:

1. N3 nodal disease according to AJCC guidelines
2. Retropharyngeal nodal involvement
3. Trismus
4. Second primary head and neck tumor unless it is/was a basal or squamous cell skin cancer
5. Prior surgery, chemotherapy, biologic or radiotherapy for a head or neck malignancy
6. Concurrent investigational agent or intervention (within 90 days of screening visit)
7. History of allergic reactions attributed to compounds of similar chemical or biologic composition to docetaxol, cisplatin, 5- fluorouracil, or carboplatin.
8. History of severe hypersensitivity reaction to drugs formulated with polysorbate 80
9. Breastfeeding women
10. Pre-existing peripheral neuropathy grade > 3
11. Evidence of distant metastatic disease
12. Unknown primary site
13. Prior or concurrent malignancies (excluding adequately treated basal or squamous cell skin cancer, in situ cervical cancer, stage I or II cancer from which the subject has been in complete remission for at least 12 months (excluding head and neck), any cancer from which the subject has been cancer free for 5 years)
14. History of allergies to any of the pre-medications.
15. Investigator consideration based upon screening interview and/or procedures
16. Evidence of bone invasion/destruction
17. Uncontrolled intercurrent illness including ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
18. Pregnant women
19. History of HIV, hepatitis B, hepatitis C, or delta antigen
20. Known allergy to India Ink or methylene blue

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Rate of pathologic complete response | 42 months
  To assess the rate of pathologic complete response of subjects (based on analysis of the surgical specimen), in both the primary site as well as the lymph nodes, with resectable stage III-IV squamous cell carcinoma of the oropharynx treated with TPF induction chemotherapy followed by conservation (organ preservation) surgery for clinically complete responders

SECONDARY OUTCOMES:
2 year overall survival | 42 months
  To assess the 2 year overall survival of subjects with resectable stage III-IV squamous cell carcinoma of the oropharynx treated with TPF induction chemotherapy followed by chemoradiation for clinically incomplete responders.
Clinical complete response | 42 months
  To report the rate of clinical complete response of the local population following TPF induction chemotherapy
2 year disease-free survival | 42 months
  To assess the 2 year disease-free survival of both subject groups
Quality of life | 42 months
  Change in quality of life status at end of treatment, 1 year, and 2 year relative to baseline
Incidence of HPV and EGFR positivity | 42 months
  To assess the incidence in both subject groups
K-ras mutational analysis | 42 months
  To assess the incidence in both subject groups

CONTACTS AND LOCATIONS:
Overall Officials: K. T. Robbins, M.D., Principal Investigator — Southern Illinois University School of Medicine; Krishna Rao, M.D., Ph.D., Principal Investigator — Southern Illinois University School of Medicine
Locations (1):
- Southern Illinois University School of Medicine, Springfield, Illinois, United States

REFERENCES:
- [Background] Robbins KT, Howell SB, Williams JS. Intra-arterial chemotherapy for head and neck cancer: is there a verdict? Cancer. 2010 May 1;116(9):2068-70. doi: 10.1002/cncr.24930. No abstract available. PMID 20186833
- [Background] Malone J, Robbins KT. Neck dissection after chemoradiation for carcinoma of the upper aerodigestive tract: indications and complications. Curr Opin Otolaryngol Head Neck Surg. 2010 Apr;18(2):89-94. doi: 10.1097/MOO.0b013e32833693e7. PMID 20125024
- [Background] Malone JP, Gerberi MA, Vasireddy S, Hughes LF, Rao K, Shevlin B, Kuhn M, Collette D, Tennenhouse J, Robbins KT. Early prediction of response to chemoradiotherapy for head and neck cancer: reliability of restaging with combined positron emission tomography and computed tomography. Arch Otolaryngol Head Neck Surg. 2009 Nov;135(11):1119-25. doi: 10.1001/archoto.2009.152. PMID 19917925
- [Background] Rogers LQ, Rao K, Malone J, Kandula P, Ronen O, Markwell SJ, Courneya KS, Robbins KT. Factors associated with quality of life in outpatients with head and neck cancer 6 months after diagnosis. Head Neck. 2009 Sep;31(9):1207-14. doi: 10.1002/hed.21084. PMID 19360748
- [Background] Robbins KT, Homma A. Intra-arterial chemotherapy for head and neck cancer: experiences from three continents. Surg Oncol Clin N Am. 2008 Oct;17(4):919-33, xi. doi: 10.1016/j.soc.2008.04.015. PMID 18722926